CLINICAL TRIAL: NCT01964521
Title: An Open, Non-comparative, Multi-centre Post Marketing Clinical Follow-up (PMCF) Investigation to Evaluate Performance and Safety on Diabetic Foot Ulcer, DFU, When Using Mepilex Transfer Ag as Intended
Brief Title: TITLE: An Open, Non-comparative, Multi-centre Post Marketing Clinical Follow-up (PMCF) Investigation to Evaluate Performance and Safety on Diabetic Foot Ulcer, DFU, When Using Mepilex Transfer Ag as Intended
Acronym: MxT Ag 05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxT Ag 05
Record Dates: First submitted 2013-09-30; First posted 2013-10-17 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2014-02

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepilex Transfer Ag (Experimental): Mepilex Transfer Ag is a transfer dressing designed for low to high exuding wounds and used to prevent microbial growth. It is worn for up to two weeks at a time.
  Interventions: Device: Mepilex Transfer Ag

INTERVENTIONS:
Device: Mepilex Transfer Ag — A soft silicone wound contact layer that absorbs and transfers exudate, maintains a moist wound healing environment and has antimicrobial properties.

SUMMARY:
An open, non-comparative, multi-centre post marketing clinical follow-up, PMCF, investigation to evaluate performance and safety on diabetic foot ulcer, dfu, when using mepilex transfer Ag as intended.

DETAILED DESCRIPTION:
Approximately 25-30 subjects from two to three centers will be evaluated provided they fulfill the inclusion criteria and none of the exclusion criteria and gives a signed and dated consent.

Subjects to be included were to suffer from a DFU and being in need of anti-microbial wound dressing.

Dressing changes were to performed according to the local clinical routine (usually 3 times/week), evaluated during a total treatment period of maximum 4 weeks including weekly visits when assessments were being done. A record (dressing log) for Mepilex Transfer Ag and outer layers were to be filled in at every dressing change.

Photos taken directly upon dressing removal and after cleansing /debridement were to be collected to visually follow the ulcers status.

At each visit the investigators/nurse and subjects opinion (using an evaluation form) were to be asked for questions considering the use of Mepilex Transfer Ag. Pain before, during and after removal will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Both gender>=18 years old
2. Subjects with type 1 or 2 diabetes mellitus
3. Two of the signs of infection must be present and recorded (redness, heat, oedema, pain, increased exudates amount, deteriorating wound, fever, odour)
4. Ulcer localization; below the ankle
5. Signed Informed Consent

Exclusion Criteria:

1. Dry wound
2. Known allergy/hypersensitivity to the dressing
3. Treated with other Silver dressing on the ulcer target within 1 week prior to this investigation
4. Subjects who will have problems following the clinical investigation plan
5. Subjects enrolled in the investigation already
6. Subjects included in other ongoing clinical investigation at present or during the past 30 days. Subjects participating in a clinical sample investigation might be enrolled in the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ketan Dhatariya, Doctor, Principal Investigator — Norfolk & Norwich University Hospitals NHS foundation
Locations (2):
- United Kingdom (2):
  - The Norfolk & Norwich University Hospitals NHS foundation, Norwich, Colney Lane
  - The Rotherham NHS Foundation Trust, Rotherham

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mepilex Transfer Ag
Started | 24
Completed | 20
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Adult subjects with diabetic foot ulcers
Groups:
- Mepilex Transfer Ag: An open, non-comparative study.
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Changes in Signs and Symptoms of Local Infection
Description: Evaluation of signs of infection (exudate) from baseline
Time Frame: 4 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Mepilex Transfer Ag
Number analyzed (Participants) | 24
Participants
  Week 1 Exudate amount - worsening compared to base | 2
  Week 2 Exudate amount - worsening compared to base | 1
  Week 4 Exudate amount - worsening compared to base | 0

2. Secondary Outcome: Levels of Pain in Connection to Dressing Changes.
Description: Levels of pain measured by VAS, visual analog scale. 1 to 100 mm, 1= low pain, 100= worse pain.
Time Frame: 4 weeks
Population: For some patients pain assessment was not performed at all predefined timepoints. Therefore some data were not collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pain by Visual Analogue Scale, LOCF: Levels of pain in connection to dressing changes.
Arm/Group | Pain by Visual Analogue Scale, LOCF
Number analyzed (Participants) | 24
units on a scale
  Baseline | 16 (24.4)
  Week 1: number analyzed (Participants) | 23
  Week 1 | 7.2 (14.3)
  Week 2 | 3.5 (4.9)
  Week 3: number analyzed (Participants) | 23
  Week 3 | 4.7 (9.8)
  Week 4: number analyzed (Participants) | 21
  Week 4 | 3.0 (4.1)

ADVERSE EVENTS:
Arm/Group | Mepilex Transfer Ag
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Transfer Ag (N=24)
pulmonary embolism (General disorders) | 1 (1)
psuedo-gout of wrist (General disorders) | 1 (1)
wound infection (Infections and infestations) | 3 (3)
Wound deterioration (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Transfer Ag (N=24)
ankle pain (General disorders) | 1 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less